CLINICAL TRIAL: NCT01946438
Title: Safety and Immunogenicity Among Adults of Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose Influenza Virus Vaccines, 2013-2014 Formulations
Brief Title: Study of Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose Influenza Virus Vaccines in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GRC52; U1111-1127-7587 (Other: WHO)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation),; Fluzone® Intradermal, Influenza Virus Vaccine (2013-2014 formulation),; Fluzone® High-Dose, Influenza Virus Vaccine (2013-2014 formulation)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) (Experimental): Participants age 18 to < 65 years randomized to receive a dose of Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation)
  Interventions: Biological: Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation),
- Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) (Experimental): Participants age 18 to < 65 years randomized to receive a dose of Fluzone® Intradermal, Influenza Virus Vaccine (2013-2014 formulation)
  Interventions: Biological: Fluzone® Intradermal, Influenza Virus Vaccine (2013-2014 formulation),
- Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) (Experimental): Participants age ≥ 65 years randomized to receive a dose of Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation)
  Interventions: Biological: Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation),
- Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4) (Experimental): Participants age ≥ 65 years randomized to receive a dose of Fluzone® High-Dose, Influenza Virus Vaccine (2013-2014 formulation)
  Interventions: Biological: Fluzone® High-Dose, Influenza Virus Vaccine (2013-2014 formulation)

INTERVENTIONS:
Biological: Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation), — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent, Influenza Virus Vaccine
  Arms: Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1)
Biological: Fluzone® Intradermal, Influenza Virus Vaccine (2013-2014 formulation), — 0.1 mL, Intradermal
  Other Names: Fluzone® Intradermal, Influenza Virus Vaccine
  Arms: Adult Fluzone® Intradermal, Influenza Vaccine (Group 2)
Biological: Fluzone® Quadrivalent, Influenza Virus Vaccine (2013-2014 formulation), — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent, Influenza Virus Vaccine
  Arms: Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3)
Biological: Fluzone® High-Dose, Influenza Virus Vaccine (2013-2014 formulation) — 0.5 mL, Intramuscular
  Other Names: Fluzone® High-Dose, Influenza Virus Vaccine
  Arms: Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)

SUMMARY:
The aim of the study is describe the safety and immunogenicity of Fluzone Quadrivalent and Fluzone Intradermal vaccines in adults 18 to < 65 years of age, and to describe the safety and immunogenicity of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.

Primary Objective:

* To describe the safety of the 2013-2014 formulations of Fluzone Quadrivalent and Fluzone Intradermal vaccines in adults 18 to < 65 years of age and the safety of the 2013-2014 formulations of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.

Observational objectives:

* To describe the immunogenicity of the 2013-2014 formulations of Fluzone Quadrivalent and Fluzone Intradermal vaccines in adults 18 to < 65 years of age and the immunogenicity of the 2013-2014 formulations of Fluzone Quadrivalent and Fluzone High-Dose vaccines in adults ≥ 65 years of age.
* To evaluate the compliance, in terms of immunogenicity, of each study vaccine (Fluzone Quadrivalent, Fluzone Intradermal, and Fluzone High-Dose) in the applicable age group with the historical requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96.
* To submit sera from selected subjects to the Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
Participants 18 to < 65 years of age on enrollment will be randomized to receive either Fluzone Quadrivalent or Fluzone Intradermal vaccine. Participants ≥ 65 years of age at enrollment will be randomized to receive either Fluzone Quadrivalent or Fluzone High-Dose vaccine.

Solicited adverse event (AE) information will be collected for 7 days after each vaccination, unsolicited AE and Serious adverse event information will be collected from Visit 1 to Visit 2. Total duration of participation in the study is approximately 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Prior vaccination with any 2013-2014 formulation of influenza vaccine
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent, Fluzone Intradermal, or Fluzone High-Dose vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, as reported by the subject
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 100.4°F]) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Santa Rosa, California
  - Council Bluffs, Iowa
  - Metairie, Louisiana
  - Cincinnati, Ohio

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 16 to 24 September 2013 at 4 clinic centers in the United States.
Pre-assignment Details: A total of 208 participants who met all of the inclusion and none of the exclusion criteria were enrolled and vaccinated in the study.
Groups:
- Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1): Participants age 18 to < 65 years who received a 0.5 mL dose of Fluzone® Quadrivalent, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
- Adult Fluzone® Intradermal, Influenza Vaccine (Group 2): Participants age 18 to < 65 years who received a 0.1 mL dose of Fluzone® Intradermal, Influenza Virus Vaccine intradermally (2013-2014 formulation)
- Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3): Participants age ≥ 65 years who received a 0.5 mL dose of Fluzone® Quadrivalent, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
- Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4): Participants age ≥ 65 years who received a 0.5 mL dose of Fluzone® High-Dose, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
Period: Overall Study
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Started | 52 | 52 | 52 | 52
Completed | 50 | 52 | 51 | 51
Not Completed | 2 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Serious Adverse event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Elderly Fluzone® High Dose, Influenza Vaccine (Group 4): Participants age ≥ 65 years who received a 0.5 mL dose of Fluzone® High Dose, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
- Total: Total of all reporting groups
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High Dose, Influenza Vaccine (Group 4) | Total
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 0 | 0 | 104
  >=65 years | 0 | 0 | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (15.2) | 46.9 (14.7) | 71.5 (4.7) | 72.6 (5.2) | 58.75 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 32 | 33 | 128
  Male | 18 | 23 | 20 | 19 | 80
Region of Enrollment [Number; unit: Participants]
  United States | 52 | 52 | 52 | 52 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection-Site and Solicited Systemic Reactions Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Fluzone® Intradermal, or Fluzone® High-Dose Vaccine.
Description: Solicited injection-site reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering. Grade 3: Pain, Significant, prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis, >100 mm; Fever, ≥102.1°F; Headache, Malaise, Myalgia, and Shivering, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 21 post-vaccination
Population: Solicited injection-site reactions and systemic reactions were assessed using the Safety Analysis Set, which includes all persons who received at least one dose of study vaccine.
Measure: Number; unit: Participants
Groups:
- Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1): Participants age 18 to < 65 years who received a dose of Fluzone® Quadrivalent, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
- Adult Fluzone® Intradermal, Influenza Vaccine (Group 2): Participants age 18 to < 65 years who received a dose of Fluzone® Intradermal, Influenza Virus Vaccine intradermally (2013-2014 formulation)
- Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3): Participants age ≥ 65 years who received a dose of Fluzone® Quadrivalent, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
- Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4): Participants age ≥ 65 years who received a dose of Fluzone® High-Dose, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Number analyzed (Participants) | 52 | 52 | 52 | 52
Participants
  Injection-site pain (N = 52, 52, 52, 52) | 27 | 30 [0 to 0] | 10 [0 to 0] | 21 [0 to 0]
  Grade 3 Injection-site pain (N = 52, 52, 52, 52) | 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection-ste erythema (N=52,52,52,51) | 0 | 15 [0 to 0] | 0 [0 to 0] | 2 [0 to 0]
  Grade 3 Injection-site erythema (N =52, 52,52, 51) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection-site swelling (N = 51, 52, 52, 51) | 1 | 2 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Grade 3 Injection-site swelling (N = 51,52,52,51) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection-site induration (N = 51, 52, 52, 51) | 1 | 4 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Injection-site induration (N= 51,52,52,51) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection-site ecchymosis (N = 51, 52, 52, 51) | 0 | 2 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Injection-site ecchymosis (N= 51,52,52,51) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Fever (N = 52, 52, 52, 52) | 0 | 0 [0 to 0] | 1 [0 to 0] | 2 [0 to 0]
  Grade 3 Fever (N = 52, 52, 52, 52) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Headache (N = 52, 52, 52, 51) | 13 | 8 [0 to 0] | 5 [0 to 0] | 8 [0 to 0]
  Grade 3 Headache (N = 52, 52, 52, 51) | 1 | 1 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Malaise (N = 52, 52, 52, 52) | 11 | 12 [0 to 0] | 2 [0 to 0] | 8 [0 to 0]
  Grade 3 Malaise (N = 52, 52, 52, 52) | 1 | 1 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Myalgia (N = 52, 52, 52, 51) | 13 | 16 [0 to 0] | 6 [0 to 0] | 10 [0 to 0]
  Grade 3 Myalgia (N = 52, 52, 52, 51) | 2 | 1 [0 to 0] | 1 [0 to 0] | 1 [0 to 0]
  Shivering (N = 52, 52, 52, 51) | 3 | 2 [0 to 0] | 2 [0 to 0] | 4 [0 to 0]
  Grade 3 Shivering (N = 52, 52, 52, 51) | 1 | 0 [0 to 0] | 0 [0 to 0] | 3 [0 to 0]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies to the Antigens Contained in the 2013-2014 Formulation of Fluzone® Quadrivalent, Fluzone® Intradermal, or Fluzone® High-Dose Vaccine Before and Following Vaccination With the Respective Vaccine
Description: Influenza virus antibodies were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 21 after vaccination
Population: Geometric mean titers of antibodies against the hemagglutinin (HA) antigens were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1): Participants age 18 to < 65 years who received a dose of Fluzone® Quadrivalent, Influenza Vaccine 2013-2014 formulation
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Number analyzed (Participants) | 49 | 52 | 51 | 51
Titers
  A/H1N1 (pre-vaccination) | 82.3 [48.0 to 141] | 74.3 [46.3 to 119] | 54.7 [36.9 to 81.1] | 91.0 [60.7 to 136]
  A/H1N1 (post-vaccination) | 514 [366 to 722] | 471 [332 to 669] | 163 [119 to 224] | 345 [255 to 467]
  A/H3N2 (pre-vaccination) | 77.2 [45.2 to 132] | 128 [81.2 to 203] | 185 [128 to 267] | 104 [67.7 to 159]
  A/H3N2 (post-vaccination) | 563 [399 to 796] | 531 [396 to 712] | 449 [344 to 587] | 636 [464 to 871]
  B (Yamagata; pre-vaccination) | 34.2 [23.3 to 50.4] | 38.2 [26.7 to 54.6] | 32.4 [24.4 to 43.1] | 36.1 [28.2 to 46.3]
  B (Yamagata; post-vaccination) | 142 [105 to 192] | 147 [110 to 196] | 67.5 [55.3 to 82.4] | 122 [98.5 to 151]
  B (Victoria; pre-vaccination) | 24.7 [17.6 to 34.7] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group | 34.2 [25.8 to 45.5] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group
  B (Victoria; post-vaccination) | 134 [96.6 to 186] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group | 67.5 [52.7 to 86.4] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group

3. Secondary Outcome: Number of Participants With Seroprotection Before and Following Vaccination With the 2013-2014 Formulation of Fluzone® Quadrivalent, Fluzone® Intradermal, or Fluzone® High-Dose Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Seroprotection was defined as a titer of ≥40 (1/dilution).
Time Frame: Day 0 (pre-vaccination) and Day 21 after vaccination
Population: Seroprotection against the hemagglutinin antigens were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- Elderly Fluzone® High Dose, Influenza Vaccine (Group 4): Participants age ≥ 65 years who received a dose of Fluzone® High-Dose, Influenza Virus Vaccine intramuscularly (2013-2014 formulation)
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High Dose, Influenza Vaccine (Group 4)
Number analyzed (Participants) | 49 | 52 | 51 | 51
Participants
  A/H1N1 (pre-vaccination) | 34 | 36 [0 to 0] | 32 [0 to 0] | 39 [0 to 0]
  A/H1N1 (post-vaccination) | 47 | 52 [0 to 0] | 47 [0 to 0] | 51 [0 to 0]
  A/H3N2 (pre-vaccination) | 33 | 41 [0 to 0] | 47 [0 to 0] | 41 [0 to 0]
  A/H3N2 (post-vaccination) | 48 | 52 [0 to 0] | 50 [0 to 0] | 51 [0 to 0]
  B (Yamagata; pre-vaccination) | 28 | 31 [0 to 0] | 26 [0 to 0] | 29 [0 to 0]
  B (Yamagata; post-vaccination) | 44 | 49 [0 to 0] | 45 [0 to 0] | 50 [0 to 0]
  B (Victoria; pre-vaccination) | 23 | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group | 32 [0 to 0] | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group
  B (Victoria; post-vaccination) | 44 | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group | 42 [0 to 0] | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group

4. Secondary Outcome: Number of Participants Achieving Seroconversion Following Vaccination With the 2013-2014 Formulations of Fluzone® Quadrivalent, Fluzone® Intradermal, or Fluzone® High-Dose Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and a ≥ 4-fold increase in titer after vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 21 after vaccination
Population: Seroconversion against the hemagglutinin antigens contained in the vaccine were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Number analyzed (Participants) | 49 | 52 | 51 | 51
Participants
  A/H1N1 | 23 | 26 [0 to 0] | 17 [0 to 0] | 25 [0 to 0]
  A/H3N2 | 27 | 19 [0 to 0] | 15 [0 to 0] | 33 [0 to 0]
  B (Yamagata) | 19 | 18 [0 to 0] | 5 [0 to 0] | 21 [0 to 0]
  B Victoria | 25 | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group | 9 [0 to 0] | NA [0 to 0] — B (Victoria) antigen was not in the vaccine administered to this group

5. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Antibodies to Antigens Contained in the 2013-2014 Formulation of Fluzone® Quadrivalent, Fluzone® Intradermal, or Fluzone® High-Dose Vaccine Following Vaccination With the Respective Vaccine
Description: Influenza virus antibodies were measured using an HAI assay. Geometric mean titer ratios are the geometric means of the individual post-vaccination/pre-vaccination titer ratios for each hemagglutinin antigen contained in the vaccines.
Time Frame: Day 21 after vaccination
Population: Geometric mean titer ratios against each hemagglutinin antigen were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Number analyzed (Participants) | 49 | 52 | 51 | 51
Titer Ratio
  A/H1N1 | 5.58 [3.29 to 9.44] | 5.77 [3.33 to 10.0] | 2.89 [2.10 to 3.97] | 3.66 [2.78 to 4.83]
  A/H3N2 | 6.42 [4.22 to 9.79] | 3.92 [2.62 to 5.87] | 2.40 [1.81 to 3.19] | 6.10 [4.12 to 9.03]
  B (Yamagata) | 3.62 [2.56 to 5.12] | 3.50 [2.36 to 5.18] | 1.95 [1.64 to 2.31] | 3.28 [2.58 to 4.18]
  B (Victoria) | 4.74 [3.23 to 6.95] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group | 1.86 [1.55 to 2.22] | NA [NA to NA] — B (Victoria) antigen was not in the vaccine administered to this group

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 21 after vaccination.
Arm/Group | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4)
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52 | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 27/52 | 30/52 | 10/52 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) (N=52) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) (N=52) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) (N=52) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4) (N=52)
Device failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Adult Fluzone® Quadrivalent, Influenza Vaccine (Group 1) (N=52) | Adult Fluzone® Intradermal, Influenza Vaccine (Group 2) (N=52) | Elderly Fluzone® Quadrivalent, Influenza Vaccine (Group 3) (N=52) | Elderly Fluzone® High-Dose, Influenza Vaccine (Group 4) (N=52)
Injection-site pain (General disorders) | 27 (27) | 30 (30) | 10 (10) | 21 (21)
Injection-site erythema (General disorders) | 0 (0) | 15 (15) | 0 (0) | 2/51 (2)
Injection-site induration (General disorders) | 1/51 (1) | 4 (4) | 0 (0) | 0/51 (0)
Headache (Nervous system disorders) | 13 (13) | 8 (8) | 5 (5) | 8/51 (8)
Malaise (General disorders) | 11 (11) | 12 (12) | 2 (2) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 16 (16) | 6 (6) | 10/51 (10)
Shivering (General disorders) | 3 (3) | 2 (2) | 2 (2) | 4/51 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications